CLINICAL TRIAL: NCT01650038
Title: Transplantation of Faeces in Ulcerative Colitis; Restoring Nature's Homeostasis.
Acronym: TURN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, C.Y. Ponsioen, MD PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: METC 2011_005
Record Dates: First submitted 2012-07-18; First posted 2012-07-26 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Ulcerative Colitis
Keywords: faecal transplantation; ulcerative colitis; inflammatory bowel disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Therapeutics; Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- faecal transplantation; donor faeces (Active Comparator): 2 times treatment with faecal transplantation: faeces from a healthy donor processed for duodenal tube infusion. after bowel lavage with macrogol.
  Interventions: Other: treatment with faecal transplantation (donor faeces)
- faecal transplantation; placebo (Placebo Comparator): 2 times treatment with (own) faecal transplantation: faeces from the patient processed for duodenal tube infusion. after bowel lavage with macrogol.
  Interventions: Other: treatment with faecal transplantation (own faeces)

INTERVENTIONS:
Other: treatment with faecal transplantation (donor faeces) — faecal transplantation
  Arms: faecal transplantation; donor faeces
Other: treatment with faecal transplantation (own faeces) — faecal transplantation
  Arms: faecal transplantation; placebo

SUMMARY:
Ulcerative colitis (UC) is a chronic inflammatory bowel disease (IBD) of the colon. Complaints such as abdominal pain, cramps and bloody diarrhoea usually start in early adulthood and lead to life-long substantial morbidity. There is no medical treatment available that meets the desired criteria of high efficacy versus low adverse effects. The current prevailing hypothesis regarding the cause of UC states that the pathogenesis involves an inappropriate and ongoing activation of the mucosal immune system driven by the intestinal microbiota in a genetically predisposed individual. Systematic investigation into the effect of correcting the dysbiosis in ulcerative colitis patients has never been performed. The most radical way to restore the presumably disturbed natural homeostasis in UC is to perform faecal transplantation from a healthy donor. In this trial the potential beneficial effects of restoring microbial homeostasis by faecal transplantation through a duodenal tube will be studied in a phase II randomised placebo controlled design.

Endpoints are clinical remission and reduction of endoscopic inflammation after 12 weeks (primary), as well as time to recurrence, intra individual changes in faecal samples and mucosal biopsies. Follow up is 12 months.

DETAILED DESCRIPTION:
treatment with faecal transplantation from a healthy donor in active ulcerative colitis patients. In this trial the potential beneficial effects of restoring microbial homeostasis by faecal transplantation through a duodenal tube will be studied in a phase II randomised placebo controlled design.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Ability to give informed consent
* Established ulcerative colitis with known involvement of the left colon according to the Lennard-Jones criteria
* SCCAI of 4 > < 11
* Endoscopic Mayo score of > 1
* Stable dose of thiopurines in preceding 8 weeks
* Stable dose of corticosteroids and 5-ASA in preceding 2 weeks

Exclusion Criteria:

* Condition leading to profound immunosuppression
* Anti-TNF treatment in preceding 2 months
* Cyclosporine treatment in preceding 4 weeks
* Use of Methotrexate in preceding 2 months
* Prednisolone dose > 10 mg
* Life expectancy < 12 months
* Use of systemic antibiotics in preceding 6 weeks
* Use of probiotic treatment in preceding 6 weeks
* Positive stool cultures for common enteric pathogens (Salmonella, Shigella, Yersinia, Campylobacter, enteropathogenic e coli)
* Positive faecal PCR-test (positive PCR means: > 1 of the following viruses is present) for: Rotavirus, Norovirus, Enterovirus, Parechovirus Sapovirus, Adenovirus 40/41/52. Astrovirus.
* Pregnancy or women who give breastfeeding
* Vasopressive medication, icu stay

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-05; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
co-primary endpoint of clinical remission, as well as reduction of Mayo endoscopic inflammation score | at 12 weeks after treatment.
  * clinical remission = questionnaire: SCCAI 2 or lower
  * reduction of Mayo endoscopic inflammation score= decrement of 1 or more as assessed by sigmoidoscopy

SECONDARY OUTCOMES:
Simple clinical colitis activity index (SCCAI) score reduction | time: 6 weeks after treatment
Frequency of bowel movements | start at baseline up to 6 weeks after treatment
Time to recurrence | from timepoint 12 weeks after treatment up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: C Ponsioen, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic_Medical_Center, Amsterdam, Netherlands

REFERENCES:
- [Derived] Rossen NG, Fuentes S, van der Spek MJ, Tijssen JG, Hartman JH, Duflou A, Lowenberg M, van den Brink GR, Mathus-Vliegen EM, de Vos WM, Zoetendal EG, D'Haens GR, Ponsioen CY. Findings From a Randomized Controlled Trial of Fecal Transplantation for Patients With Ulcerative Colitis. Gastroenterology. 2015 Jul;149(1):110-118.e4. doi: 10.1053/j.gastro.2015.03.045. Epub 2015 Mar 30. PMID 25836986